CLINICAL TRIAL: NCT04492293
Title: A Phase 2, Multicenter, Single Arm, Open-lable Study of ICP-192 in Subjects With Surgically Unresectable or Metastatic Bladder Urothelial Cancer With FGFR Genetic Aberrations.
Brief Title: An Efficacy and Safety Study of ICP-192 in Subjects With Bladder Urothelial Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00302
Record Dates: First submitted 2020-07-23; First posted 2020-07-30 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Bladder Urothelial Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICP-192 (Experimental): ICP-192
  Interventions: Drug: ICP-192

INTERVENTIONS:
Drug: ICP-192 — ICP-192 is a white, round, uncoated table

SUMMARY:
This is a phase 2, multicenter, single arm, open-lable study of ICP-192. The purpose of this study is to evaluate efficacy of ICP-192 in subjects with surgically unresectable or metastatic bladder urothelial cancer.

DETAILED DESCRIPTION:
bladder urothelial cancer

ELIGIBILITY:
Inclusion criteria：

1. Signed the ICF and Age ≥ 18 years old, either sex.
2. ECOG ≤ 1.
3. Life expectancy of at least 3 months.
4. Histologically confirmed unresectable or metastatic bladder urothelial cancinoma.
5. At least one measurable lesion as the target lesion at screening assessed according to RECIST V1.1

Exclusion Criteria:

1. Prior treatment with selective FGFR inhibitors or FGFR antibodies.
2. Any corneal or retinal abnormalities that may result in an increased risk of ocular toxicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2020-05-27 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR | From the time of first dose until objective disease progression, an average of 6 months
  Objective Response Rate

SECONDARY OUTCOMES:
DOR | From the time of first dose until objective disease progression, an average of 6 months
  Duration of response
DCR | From the time of first dose until objective disease progression, an average of 6 months
  Disease Control Rate
PFS | From the time of first dose until objective disease progression, an average of 6 months
  Progression Free Survival
OS | From the time of first dose until objective disease progression, an average of 1 months
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (22):
- China (22):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The fifth Medical Center of People's Liberation Army General Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Union Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - The First Hospital of JiLin University, Jilin, Jilin
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Shandong University Qilu Hospital, Jinan, Shandong
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejing